CLINICAL TRIAL: NCT03499405
Title: CIN001-HeadStart Navigator Intervention
Brief Title: Head Start Family Navigator Intervention
Acronym: HeadStartNav
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Office of Head Start (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CIN001-HeadStart Navigator Int
Record Dates: First submitted 2017-12-19; First posted 2018-04-17 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Developmental Delay
Keywords: development and health disparities and navigation
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Intervention Model Description: Intervention group will have access to a culturally matched family navigator, control group will not have access to a culturally matched family navigator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention group will receive a family navigator intervention from a culturally matched family navigator.
  Interventions: Behavioral: Family Navigator Intervention
- Control group (No Intervention): Control group will not receive a family navigator intervention from a culturally matched family navigator.

INTERVENTIONS:
Behavioral: Family Navigator Intervention — Caregivers will be paired with a culturally matched family navigator.
  Arms: Intervention group

SUMMARY:
Headstart (HS) is an early childhood education program for low-income children. Preliminary analyses of Hamilton County HS preschoolers with developmental concerns identified 26% with "severe concern" necessitating developmental testing, and only 47% followed-through when some developmental concern was identified. Those less likely to follow-through were African American or Hispanic, lived in larger families, or had asthma. Cultural and economic factors are known barriers to earlier diagnosis of children with developmental disabilities (DD) among African American, Hispanic and low-income children. Given that HS children are low-income and culturally diverse, preschoolers are likely to face barriers to early identification of DD and subsequently kindergarten readiness. Patient navigator programs are effective interventions for vulnerable populations to improve health care access, increase treatment adherence, enhance trust in health care systems, and reduce health care costs. A family (FN) intervention that is culturally-adapted to promote caregiver follow-through, and undergirded by HS's mission of kindergarten success may effectively increase caregiver adherence to developmental testing. The goal of this study is to develop and pilot test a FN intervention in HS that is executed by peer-to-peer navigators to improve adherence with developmental testing in high-risk preschoolers.

DETAILED DESCRIPTION:
Headstart (HS) is a pipeline for early school success for low-income children aged 3-5 years, and provides health promotion services such as developmental monitoring to promote school readiness. In 2014-2015 Hamilton County Headstart (HCHS) identified 968 of 2987 preschoolers (32%) with developmental concern, with 251 (26%) identified as "severe concern" necessitating developmental testing. Yet, follow-through with testing did not occur for 53 high-risk preschoolers (21%), and only 451 (47%) followed-through when some developmental concern was identified. Those less likely to follow-through were African American or Hispanic, lived in families of 3 or more, or had asthma. That race and ethnicity predict insufficient follow-through is not surprising; cultural and economic factors are known barriers to earlier diagnosis of children with developmental disabilities (DD), resulting in 2 year lags in obtaining DD diagnoses among African American, Hispanic and low-income children and placing them at risk for worse long-term prognosis. Diagnostic disparities are also grounded in the social factors of poorer health care access, caregiver distrust of health systems, knowledge deficits, and stigma about disability. One mechanism thought to contribute to the diagnostic delays is caregiver postponement in obtaining developmental assessments due to these collective factors. Given that all HS children are low-income and a majority are African American or Hispanic, HS preschoolers are likely to face barriers to early identification of DD and subsequently kindergarten readiness. An intervention that addresses the salient barriers to developmental assessment for HS preschoolers could advance pre-academic abilities and promote access to earlier recognition and treatment of DD, leading to improved health outcomes.

Patient navigator programs have been effective interventions for vulnerable populations to improve health care access, increase treatment adherence, enhance trust in health care systems, and reduce health care costs. Despite these findings, investigations into peer-based navigation interventions for families of children with inferior health outcomes have mostly been program evaluations or unpublished clinical trials. A promising study in Developmental and Behavioral Pediatrics (DBP) on family navigators (FN) for children referred from primary care for evaluation of DD is examining family quality of life outcomes prior to and after DD diagnoses, and has shown preliminary success in developing and training FNs. A FN intervention that is culturally-adapted to promote caregiver follow-through, and undergirded by HS's mission of kindergarten readiness may effectively increase caregiver adherence to developmental testing in HS. The goal of this study is to refine and pilot test a FN intervention that is informed by HS caregivers, staff and primary care providers (PCP), grounded in the HS community, and executed by peer-to-peer navigators to improve adherence with developmental testing in high-risk preschoolers. This study is the final year of a research program that will focus on tailoring the elements of a community-based (Head Start (HS) Family Navigator (FN) intervention for high risk children with developmental concerns in order to improve access to developmental testing. This study will be conducted over a 1 year period with the specific aim outlined below.

The study titled: Prototype of a Head Start Navigator Intervention for Child Developmental Testing (IRB#2016-4253) was conducted to develop a community-based family navigator intervention for preschoolers identified in HS as high-risk for developmental delay. Focus groups were conducted with caregivers, teachers and primary care providers (PCPs) to understand the barriers and facilitators to follow-through with developmental testing. The prototype was tailored to the thematic focus group findings, cultural and risk factors previously identified, and results of an updated analysis of predictors of poor follow-through of developmental assessments from HCHS academic year 2015-2016 (IRB# 2016-4253). Findings confirmed that primary care and Head Start operate in silos regarding developmental screening and follow-through for at-risk children. Facilitating factors to caregiver follow-through were identified as: building relationships, increasing resource knowledge, and addressing denial/stigma of disability. Findings substantiated that caregivers needed assistance with navigating developmental testing, and valued its delivery using a peer-to-peer approach that was culturally-matched. The intervention was adapted from the crucial components necessary for a successful Family Navigator training program and delivery of the intervention including elements of frequency, duration and intensity that were also confirmed by the findings.

Materials and Methods

Study Purpose:

The study purpose is to test a community-based family navigator intervention for preschoolers identified in HS as high-risk for developmental delay. The community-based intervention will train racially/ethnically matched peer caregivers in HS as FNs. FNs from HS will guide and support caregivers to follow-through with child developmental testing. The investigators will test if a Head Start FN program is feasible, acceptable and health-promoting.

Specific Aims:

Aim 1: Pilot test a community-based FN intervention in HS that trains peer caregivers as FNs to guide and support caregivers to follow-through with child developmental testing. The investigators will test if an adapted model of a FN program that includes racially/ethnically matched peers, trained to support and guide caregivers through child developmental testing, is feasible, acceptable and health-promoting.

Key outcomes are: 1) proportion of children who complete developmental testing guided by FNs (feasibility), 2) caregiver, FN, teacher and PCP satisfaction with the intervention and its implementation (acceptability), and 3) caregivers' and FNs' knowledge of development and disparities in early DD recognition (health promotion).

Study Settings:

1. The study settings will be multiple with the primary setting being Hamilton County Head Start centers from CAA (Community Action Agency) and ESC (Educational Services Center). HS is a federally-funded program providing preschool education and kindergarten preparation. HS establishes partnerships with caregivers and communities by identifying and building on family and community strengths. Both informally and formally through parent groups and committees, caregivers are empowered to participate in HS curriculum planning and make decisions regarding their children's education. HS encompasses urban and suburban center-based programs serving income-eligible families of children 3-5 years old.
2. Additional study settings will be the caregiver's home, developmental testing sites such as primary care provider office, Cincinnati Children's Hospital Medical Center, Division of Developmental and Behavioral Pediatrics (DDBP) outpatient clinic, therapy evaluation and treatment centers (i.e. speech, occupational, physical therapies), local school, and community locations that are mutually determined between caregiver and FN.

Participants:

1. FN participants will be current, former, or pending HS parents, or a parent of a child with a developmental disability who has experience with HS, and sampled from urban and suburban HS. Eight FNs will be trained to support and guide caregivers through developmental testing, including 4 African American, 1 Caucasian and 3 bi-lingual Hispanic parents. Each FN will be assigned 1 to 5 caregivers.
2. The study sample of caregiver participants will include 32 eligible HS caregivers of preschoolers between 3 and 5 years old identified with moderate or severe developmental concerns on HS developmental screening, in order to include those at-risk before kindergarten age. Those with moderate developmental concern will have failed 2 domains on developmental screening, whereas those with severe concern have failed 3 or more domains. Those who fail 1 domain (mild concern) will be excluded since often single domain failures are due to limited early learning exposures and/or language barriers, which can be adequately addressed in HS. Half of those selected will be sampled from the moderate and half from the severe group, with 50% from urban and 50% from suburban HS centers included. Given that the demographics differ slightly in racial and ethnic make-up among the urban and suburban Head Starts, 12 African American, 2 Caucasian and 2 Hispanic caregivers will be sampled from urban HS; in suburban HS, 8 African American, 6 Caucasian and 2 Hispanic caregivers will be sampled.

Procedures:

Recruitment:

Family Navigator recruitment: Eligible FN participants will be current, former, or pending HS parents, or a parent of a child with a developmental disability who has experience with HS, and sampled from urban and suburban HS. Recruitment will occur via purposeful sampling from HS staff, parent advisory groups, and previously completed focus group participants (IRB# 2016-4253).

Caregiver recruitment: Eligible caregiver participants will be selected for the intervention and control (usual care) groups using stratified block random sampling by race, level of developmental concern and within each urban and suburban HS center. HS database will be accessed retrospectively for the intervention and control groups. Since HS developmental screening is completed within 45 days of enrollment, selection will begin once all HS screening has been completed. The investigators will abstract data on severity of concern and whether developmental referrals were completed.

Study Procedure:

The intervention includes a training and navigation component. The training and navigation components will be adapted from an existing DDBP FN program and integrated with the intervention development features from the previous prototype study. The FN training component will be built from the DDBP FN curriculum and include training in: 1) confidentiality and HIPAA, 2) safety issues and reporting concerns, 3) disparities in identification of developmental delay and importance of early developmental testing, 4) HS and primary care and other developmental services, and 5) peer mentoring skills. The training will be provided by the research team, including consultation with HS staff and the DDBP FN. Training will include 6 hours of didactic and interactive sessions in a workshop format. The navigation component will also be developed from the DDBP FN program and generally comprise the FN role of guiding and supporting caregivers in navigating the educational and health care interfaces. The primary interfaces between FN and caregiver participants can include, but are not limited to: 1) HS identification of child at-risk for developmental concern, 2) HS and PCP communication about the child's ongoing developmental concerns and the plan for further testing/treatments, and 3) results sharing. Non-English speaking caregivers will be provided a translator for on-site HS or developmental meetings as a standard of care. The FN will build a supportive relationship with the caregiver by facilitating and guiding at each of the above interfaces through in-person meetings, attending testing and results, and facilitating communication at every interface. Intermittent FN contact with caregivers between meetings may also take the form of phone calls, texts or emails, as determined by the FN/caregiver dyad. The research team will assess the FN fidelity to the intervention with focus on the FN/caregiver dyad relationship at the mid-intervention caregiver/FN encounter. Family navigation will cease at the end of the academic year, with transitions facilitated to social service or health care agencies for severe needs not fully addressed. The navigation component will comprise about 5 two-hour meetings among the FN/caregiver dyad during the academic year.

The caregiver intervention group will include those caregivers' whose children fail 2 or more developmental domains on HS screening and will be referred for usual care in Head Start, such as follow up with primary care or school district testing . The investigators will request the caregivers share the results of any follow up visits for development (ie. with primary care or school district) with the Family Navigator, and subsequently the research team. Results will be tracked until the end of the study. The control group will be assessed from the HS database retrospectively, including access to usual care (e.g. outside referral for developmental testing in school district or primary care) when identified by HS with developmental concern.

Investigator-developed questionnaires in English or Spanish on knowledge of health disparities in DD and the importance of developmental testing will be administered to FNs and caregivers pre-and-post navigator intervention. Investigator-developed questionnaires on satisfaction and implementation of the intervention will be administered to FNs, caregivers, teachers and PCP post-intervention. Teacher and PCP questionnaires will ascertain additional factors of communication of developmental concerns between Head Start and Primary Care, and the navigator interfaces with each site. Demographic information on caregiver age, race/ethnicity, language, family size, employment, income, education, and marital status will be collected from HS records. Demographics on child age, health screenings and conditions, and HS attendance will be obtained from HS records. Completion of developmental referrals will be obtained from HS database for the intervention and control groups.

Outcome Measures:

Key outcomes for this study are: 1) proportion of children who complete developmental testing guided by FNs (feasibility), 2) caregiver, FN, teacher and PCP satisfaction with the intervention and its implementation (acceptability), and 3) caregivers' and FNs' knowledge of development and disparities in early DD recognition (health promotion).

The primary outcome is the proportion of children who complete referrals for developmental testing in the intervention group relative to the control group, with the hypothesis that the FN intervention will increase caregiver completion of referrals and time to completion is less than those in the control group (feasibility). Secondary outcomes are: 1) caregiver, FN, teacher and PCP satisfaction with the intervention and implementation (acceptability) and 2) caregiver and FN knowledge of child developmental disparities (health promotion).

Data Analysis:

The sample size of 32 caregiver participants was selected because the capacity for FNs to be trained and intervene is limited to 5 families for each of the 8 navigators, as this is a new intervention within the HS setting and feasible for newly-trained FNs in a pilot study. To assess the primary outcome, the proportion of children who complete referrals for testing will be compared between caregivers who receive the intervention and those in the control group. Participants (caregivers) will be randomized to receive either the family navigator intervention or control (usual care process) groups using stratified block random sampling by race and within each center (CAA, ESC). To compare the difference in the time from referral to testing between groups, survival analyses (e.g. Cox proportional hazards modeling) will be used. Preliminary analysis of HS caregiver completion of referral (the primary outcome of our proposed study) indicated that approximately 50% of caregivers across all groups completed a referral. With 32 moderate and severe risk preschoolers per group (32 in intervention and 32 in non-intervention), using a chi-square test with 2-sided significance level set at α=0.05 the investigators will have >90% power to detect an increase of 50% to 90% of caregivers completing the referral. Secondary outcomes include the time to completion of referrals, and acceptability and knowledge of the intervention as measured by investigator-developed instruments. These analyses will provide effect sizes for investigator-development instruments, and will enable power calculations for a subsequent R21 proposal testing random allocation of a FN intervention. Costs and labor of the intervention vs. the control group will be analyzed using means and ratios of labor costs, materials, transportation, caregiver's time off work, retention and health services use to facilitate development of procedures for wider dissemination and sustainability. The aggregate of these measures will assist our evaluation of the components needed to provide a timely, coordinated approach to follow-through with developmental testing for moderate and severe at-risk preschoolers in HS. Generalizability will be constrained by the sample size and the local sample represented, with the objective at present being to conduct a pilot intervention study. Caregiver demographic characteristics will be assessed for distribution of the data using means and standard deviations or medians and ranges as appropriate to the data.

Data Storage All electronic data and data analysis results will be stored on a password-protected limited-access network drive. Names will not be associated with the participants or risk analyses data. Only the personnel directly involved in the study will have access to the data.

Risk and Benefit to Participants The study poses minimal risk and may have no direct benefit to individuals participating in the study. However this study has the potential to add to our understanding regarding the feasibility of peer-matched navigators guiding caregiver follow-through to developmental recommendations for high-risk preschoolers. Despite having no immediate and direct benefit for the study participants, participation may benefit caregivers in obtaining developmental resources for their at-risk preschooler, and may benefit FN participants by participation in resource training.

Potential Risks, Discomforts, Inconveniences, and Precautions There is minimal risk for this study. Participants include caregivers of preschoolers enrolled in HS, current or former or pending HS parents (the family navigator participants), HS teachers and primary care providers (PCPs). Caregiver participants will be sampled to represent the cultural diversity of HS parents because the investigators are seeking to understand the feasibility of a culturally-matched peer navigator intervention to increase follow-through with developmental testing. Caregivers whose primary language is Spanish will be included and interpreter services available.

For caregiver participants it is unlikely, but possible, that after consenting they may feel uncomfortable with the emotional content around their child at-risk for developmental concerns, and if this is the case, have the right to withdraw from the study at any time. It will be reinforced in the consent that participation is voluntary, and if the process is uncomfortable for the participants they may withdraw at any time. Community resources will be offered if needed. Members of the research team will comply with requests to withdraw or no longer participate.

Private space in HS will be provided for meetings between FN and caregiver participants as needed. Caregiver participant demographics will be obtained from HS database and shared only with the research team. Caregiver, FN, teacher and PCP data from questionnaires will be shared only with the research team. Control group demographics will be obtained from HS database, and shared only in aggregate form. All sources will be de-identified.

Confidentiality Loss of confidentiality or privacy is another possible risk for the participants. To reduce these risks, the FN training will include the need to protect caregiver participant confidentiality (e.g HIPPA and FERPA) and caregivers will be informed that the FN and Caregiver meetings constitute questions and answers in a dyad. Participant names will be known only to the research team, HS site coordinators and the assigned Family Navigator. Only personnel directly associated with the study will have access to the data. Participant information and study results will be reported in aggregate. Risk analyses are conducted from de-identified data in aggregate. No identifying information will be included in scientific reports, presentations, or publications.

Method to be used in Procuring Consent of Participants The research involves no more than minimal risk to the participants and will not adversely affect the rights or welfare of the participants. All Family Navigator and Caregiver participants will be fully informed and consented for their participation. The caregiver consent form will also give parental permission for their child (age 3-5) to participate in developmental testing at CCHMC. A member of the research team will review the study information and consent with the participants using lay language. The participants will be given an opportunity to ask questions about the study. Participants will be informed that they have the right to stop participating at any time. Participation is always voluntary. The participants will be given the consent to take home to make an informed and independent decision regarding whether to participate in the research. For Spanish-speaking participants, the consent will be conducted with a Spanish-speaking translator available during consent. In addition, the investigators will translate the consent form to Spanish using the CCHMC interpreter services after IRB approval. This will be certified, and submitted to the IRB.

Additionally, approximately 25% of the Family Navigator and Caregiver participants may be Latino immigrants, a vulnerable population, who may be undocumented and/or illiterate. Having the Latino participants sign their name to a consent form would have the potential for putting the immigrant participants at risk for harm about their legal status, harm from a breach of confidentiality, and they may not be able to write their name if illiterate. For these participants, only first names will be recorded and/or linked to any information that is discussed.

Data and Safety Monitoring Plan This proposal is a pilot test of a clinical trial, and as such it will be registered at www.clinicaltrials.gov. Although given the nature of the study the investigators do not expect to have serious adverse events, the investigators are prepared to address these appropriately should they occur. The PI will be available on cell phone at all times. All numbers will be provided to all participants. Adverse events will be brought to the immediate attention of the PI through the investigative team, Head Start staff or any study participants. For recruitment of participants the PI will be available on cell phone at all times. The PI will be available at all times for any questions from the family navigators or caregiver participants about any aspects of the study. Satisfaction with the intervention will be assessed at specified intervals with questionnaires given to participants and an open-ended comment section included in the questionnaire. The PI or CRC will review all data as it is collected to monitor for safety issues. The PI will be notified immediately of any safety issues. Adverse events will require a timely response to ensure the health and well-being of participants, and procedures will be reviewed to determine their potential contribution to the adverse event. Procedural changes will ensue if they are deemed to be necessary. These will be done in conjunction with the IRB and guidance from the PI's research mentors of Dr. Tanya Froehlich (DDBP) or Dr. Rita Pickler (OSU). Both are experienced as intervention researchers in adverse event monitoring and reporting. At quarterly meetings with the research mentors, and monthly meetings with the research team, the PI will review recruitment and data collection to track the meeting of study objectives. Summary reports of data will be prepared by the PI for review by the research team prior to each meeting. The mentorship team can request additional information to assist in safety monitoring. Written minutes of these meetings with summaries of adverse events will be forwarded to the IRB and NIH as part of the annual reporting process, following institutional and NIH guidelines. Determinations or recommendations for early stopping of the pilot trial by the research team (including the research mentors) will be for reasons of safety only.

ELIGIBILITY:
Inclusion Criteria:

1. FN participants will be current or former HS parents and sampled from urban and suburban HS.Eight FNs will be trained to support and guide caregivers through developmental testing, including 4 African American, 2 Caucasian and 2 bi-lingual Hispanic parents. Each FN will be assigned 1 to 4 caregivers.
2. The study sample of caregiver participants will include 32 eligible HS caregivers of preschoolers between 3 and 4 years old identified with moderate or severe developmental concerns on HS developmental screening, in order to include those at-risk before kindergarten age. Those with moderate developmental concern will have failed 2 domains on developmental screening, whereas those with severe concern have failed 3 or more domains. Those who fail 1 domain (mild concern) will be excluded since often single domain failures are due to limited early learning exposures and/or language barriers, which can be adequately addressed in HS.24,25 Half of those selected will be sampled from the moderate and half from the severe group, with 50% from urban and 50% from suburban HS centers included. Given that the demographics differ slightly in racial and ethnic make-up among the urban and suburban Head Starts, 12 African American, 2 Caucasian and 2 Hispanic caregivers will be sampled from urban HS; in suburban HS, 8 African American, 6 Caucasian and 2 Hispanic caregivers will be sampled.

Exclusion Criteria:

* For FN, not being a former head start parent.
* For caregiver, child not failing more than 2 or more domains on developmental testing.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Proportion of children who complete developmental testing guided by family navigators (feasibility). | Up to three months.
  The primary outcome is the proportion of children who complete referrals for developmental testing in the intervention group relative to the control group, with the hypothesis that the FN intervention will increase caregiver completion of referrals and time to completion is less than those in the control group (feasibility).

SECONDARY OUTCOMES:
Caregiver satisfaction with the intervention and implementation | Up to two months.
  Caregiver satisfaction with the intervention and implementation (measured using the Investigator-developed Acceptability Questionnaire). This is a 5 point Likert scale.
Family Navigator satisfaction with the intervention and implementation | Up to two months.
  Family Navigator satisfaction with the intervention and implementation (measured using the Investigator-developed Acceptability Questionnaire). This is a 5 point Likert scale.
Teacher satisfaction with the intervention and implementation | Up to two months.
  Teacher satisfaction with the intervention and implementation (measured using the Investigator-developed Acceptability Questionnaire). This is a 5 point Likert scale.
Primary Care Provider satisfaction with the intervention and implementation | Up to two months.
  Primary Care Provider satisfaction with the intervention and implementation (measured using the Investigator-developed Acceptability Questionnaire). This is a 5 point Likert scale.
Caregiver Knowledge of child developmental disparities (health promotion). | Up to two months.
  Caregiver knowledge of child developmental disparities assessed using a pre-post knowledge questionnaire. This is a 3 point scale (True, False, Don't know).
FN knowledge of child developmental disparities (health promotion). | Up to two months.
  FN knowledge of child developmental disparities assessed using a pre/post knowledge questionnaire. This is a 3 point scale (True, False, Don't know).

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smith T, Burkett K, Pickler R, Bowers K, Weber S, Trenkamp E, Heeman A, Stanton-Chapman T, Copeland K, Froehlich T. Feasibility, Acceptability, and Preliminary Effectiveness of Family Navigation for Low-income Ethnoracially Diverse Preschoolers with Developmental Concern. J Racial Ethn Health Disparities. 2025 Sep 16. doi: 10.1007/s40615-025-02556-w. Online ahead of print. PMID 40956380